CLINICAL TRIAL: NCT02030912
Title: Phase 4 Study Into the Effect of Minocycline and Amoxicillin Administration of the Prevalence of Antibiotic Resistant Bacteria and on the Indigenous Oral, Faecal, Cutaneous and Nasal Microbiotas
Brief Title: Effect of Minocycline & Amoxicillin on Antibiotic Resistant Bacteria and Indigenous Microbiotas
Acronym: ANTIRESDEV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helperby Therapeutics Ltd (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: C09040
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Antibiotic Resistant Bacteria
Keywords: The impact of a number of different types of antibiotics; The emergence and persistence of antibiotic resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 doses of amoxicillin daily for 7 days (Active Comparator): Cohort A: 3 doses of amoxicillin daily for 7 days (n=14). Follow up 12 months.
  Interventions: Drug: 3 doses of amoxicillin daily for 7 days
- 2 doses of minocycline daily for 5 days (Active Comparator): Cohort B: 2 doses of minocycline daily for five days (n=14). Follow up 12 months.
  Interventions: Drug: 2 doses of minocycline daily for five days
- 2 doses of placebo daily for 5 days (Placebo Comparator): Cohort C: 2 doses of placebo daily for five days (n=14). Follow up 12 months.
  Interventions: Other: 2 doses of placebo daily for five days

INTERVENTIONS:
Drug: 3 doses of amoxicillin daily for 7 days
  Arms: 3 doses of amoxicillin daily for 7 days
Drug: 2 doses of minocycline daily for five days
  Arms: 2 doses of minocycline daily for 5 days
Other: 2 doses of placebo daily for five days
  Arms: 2 doses of placebo daily for 5 days

SUMMARY:
A randomised, open labelled study design is selected in order to determine the emergence and persistence of antibiotic resistant bacteria in humans and on the composition of the indigenous microbiotas at various body sites. These will involve the administration to volunteers of minocycline and amoxicillin- a control group will receive a placebo. Microbiology of the skin, saliva, faecal, skin and nasal micro flora, safety and adverse events, vital signs, will be evaluated. The objectives of metagenomic analysis are:

* To identify the in vivo molecular mechanisms responsible for antibiotic resistance and its transfer in the indigenous oral and faecal microbiotas using metagenomics resistome analysis.
* To determine the impact of the use of antimicrobial agents on the oral resistome
* To determine the impact of the use of antimicrobial agents on the faecal resistome
* To determine the ecological impact of the use of antimicrobial agents on the relative abundance of phylotypes of the indigenous oral microbiota
* To determine the ecological impact of the use of antimicrobial agents on the relative abundance of phylotypes of the indigenous faecal microbiotas

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 40 years.
2. Following verbal & written information about the trial, the subject has signed & dated informed consent before any study related activity was carried out.
3. Subject legally competent and able to communicate effectively with the study personnel
4. Normal finding in the medical history and physical examination, unless the investigator considers an abnormality to be clinically irrelevant.
5. Male or female subjects who are using a medically acceptable method of contraception or of non-childbearing potential (i.e., surgically sterile-bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing or naturally postmenopausal for at least one year with a Screening FSH leve≥l 40 mIU/L). - - A negative serum pregnancy test is required at Screening for females.

Exclusion Criteria:

1. Regular use of medication, except contraceptive, vitamin tablets, treatment with antimicrobial agents within the 3 months preceding the study, Use of antibiotics for 4 weeks prior to the study drug application or use of concomitant systemic or topical antibiotics, Systemic treatment with immunosuppressive drugs e.g. cyclosporine, azathioprine or oral corticosteroids within 4 weeks prior to baseline visit (Visit 2) .
2. Participation in a trial with another investigational drug within the 3 months preceding the study
3. Present or residual gastrointestinal, renal insufficiency or hepatic disorder
4. Abnormal pathology of nasal passages
5. Any clinically significant allergy or drug intolerance
6. Active hay fever, on-going cold/flu symptoms, including rhinitis at baseline (visit 2)
7. Any medical history of renal insufficiency or hepatic disorder or other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs
8. history of hypersensitivity to beta-lactams or tetracycline
9. pregnant or breast-feeding women
10. Subjects known or suspected of not being able to comply with trial protocol (e.g. alcoholism, drug dependency, or psychological state). History of regular alcohol consumption exceeding an average weekly intake of alcohol greater than 21 units for female and 28 units for male.

    One unit is equivalent to a half-pint of beer or one measure of spirits or one glass of wine.
11. Subjects with known or suspected immunodeficiency.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percentage of resistant bacteria collected from body sites in subjects receiving minocycline/ amoxicillin compared to the baseline. | 12 Months

SECONDARY OUTCOMES:
Adverse events (AEs) will be monitored throughout the study | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd, London, London, United Kingdom